CLINICAL TRIAL: NCT01819116
Title: Tissue Oxygen Saturation During Management of the Deceased by Neurological Criteria Organ Donor as a Predictor of Number of Organs to Transplant Per Donor
Brief Title: Organ Donor Tissue Oxygen Saturation as a Predictor of Number of Organs to Transplant Per Donor
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Silvia Perez-Protto, MD, M.D., The Cleveland Clinic
Other Study IDs: 13-020
Record Dates: First submitted 2013-03-19; First posted 2013-03-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2014-03

CONDITIONS: Brain Death
Keywords: Tissue Oxygen Saturation; Management of the DNC Organ Donor
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to quantify the association between tissue oxygen saturation (StO2) during the donor management phase of the Death by Neurological Criteria (DNC) organ donor and the number of organs transplanted per donor.

DETAILED DESCRIPTION:
Specifically the study aims to:

1. Evaluate the association between StO2 level in the DNC organ donor and the number of organs transplanted per donor;
2. Evaluate whether or not tissue perfusion in the DNC organ donor population correlates with currently measured macro-hemodynamic variables during the donor management phase.
3. Assess if StO2 in the DNC organ donor is related to the number of organs with normal end-organ function, and with the number of organs predicted to be transplanted using the organ donor calculator.
4. Assess if StO2 in the DNC organ donor is related with intravenous thyroid hormone treatment.

Investigators will conduct an observational study, including 60 DNC organ donors, in Lifebanc's Donor Service Area (DSA). Investigators will monitor and record blindly the StO2 with near-infrared spectroscopy (NIRS) in the DNC organ donor from the beginning of the OPO (Organ Procurement Organization) organ donor management period until cardiac arrest in the operating room at the time of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. DNC organ donor
2. Age ≥ 15 years old
3. Weight ≥ 45 Kg

Exclusion Criteria:

1. Donor after circulatory determination of death
2. Living donor

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: DNC Organ Donor managed by Lifebanc
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of organs transplanted per donor | At 24 hours after transfering the donor to operating room.

SECONDARY OUTCOMES:
Number of organs with targeted end-organ function per donor | At the last hour at the Intensive Care Unit, before the donor is transferred to the operating room.
  Normal end-organ function definitions
  1. Kidney function: Creatinine ≤ 1.5 mg/dL, urinary output ≥ 0.5 ml/kg/h
  2. Liver function: INR <1.5, Prothrombin time: 8.4-13 seconds (or within normal range per testing lab). Bilirubin, AST, ALT within normal range per laboratory limits.
  3. Lung function: PaO2/FiO2 index ≥ 300 with PEEP ≤ 8 (oxygen challenge gas)
  4. Heart function: Normal systolic and diastolic function per echocardiogram with minimal inotropic/vasopressor support. Systolic function will be estimated by ejection fraction and/or shortening fraction on echocardiogram. Normal cardiac catheterization data if available
  5. Pancreatic function: HbA1c<6, amylase and lipase within normal range per laboratory limits.
  6. Small intestine function: lactate ≤ 2.2 mmol/L with minimal vasopressor support.
Number of organs predicted to be transplanted using organ donor calculator | At the last hour at the Intensive Care Unit, before the donor is transferred to the operating room.
Correlation of tissue oxygenation readings to macro-hemodynamic measurements | During donor management until cardiac arrest at the operating room
  Mean arterial pressure, central venous pressure, cardiac output, positive pressure variation, stroke volume variation
Variation of tissue oxygenation after thyroid hormone is initiated, titrated and/or discontinued. | During donor management until cardiac arrest at the operating room

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Perez-Protto, MD, Principal Investigator — The Cleveland Clinic; Daniel Lebovitz, MD, Study Director — Akron Children Hospital - Lifebanc; J. Steven Hata, MD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States